CLINICAL TRIAL: NCT02005471
Title: A Multicenter, Phase III, Open-Label, Randomized Study in Relapsed/Refractory Patients With Chronic Lymphocytic Leukemia to Evaluate the Benefit of Venetoclax (GDC-0199/ABT-199) Plus Rituximab Compared With Bendamustine Plus Rituximab
Brief Title: A Study to Evaluate the Benefit of Venetoclax Plus Rituximab Compared With Bendamustine Plus Rituximab in Participants With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Acronym: MURANO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO28667; 2013-002110-12 (EudraCT Number)
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; venetoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Bendamustine + Rituximab (Active Comparator): Participants will receive bendamustine 70 milligrams per meter square (mg/m^2) via intravenous (IV) infusion on Days 1 and 2 of each 28-day cycle for 6 cycles, in combination with rituximab 375 mg/m^2 via IV infusion on Day 1 of Cycle 1 followed by 500 mg/m^2 on Day 1 of Cycles 2-6.
  Interventions: Drug: Bendamustine; Drug: Rituximab
- Venetoclax + Rituximab (Experimental): Participants will be initially placed on a venetoclax 5 weeks ramp-up period, and will receive an initial dose of 20 milligrams (mg) via tablet orally once daily (QD). Then the dose will be incremented weekly up to a maximum dose of 400 mg. Participants will then continue receiving venetoclax 400 mg QD from Week 6 (Day 1 of Cycle 1 of combination therapy) onwards, as directed by the investigator, in combination with rituximab 375 mg/m^2 via IV infusion on Day 1 of Cycle 1 followed by 500 mg/m^2 on Day 1 of Cycles 2-6.
  Interventions: Drug: Venetoclax; Drug: Rituximab
- Bendamustine + Rituximab Crossover Substudy (Experimental): Participants entering the Crossover Substudy will have a 5-week venetoclax dose ramp-up period to reach the target dose of 400 mg QD. Following the venetoclax ramp-up period, Participants will receive 6 cycles of rituximab consisting of a single infusion on the first day of each 28-day cycle. Participants will continue to take their daily dose of venetoclax during the rituximab cycles. Participants who have not progressed following the completion of the 6 cycles will continue to receive venetoclax monotherapy until disease progression or for a maximum of 2 years from Cycle 1 Crossover Day 1 of the Substudy.
  Interventions: Drug: Venetoclax; Drug: Rituximab
- Venetoclax + Rituximab Re-Treatment (Experimental): Participants entering the Re-Treatment Substudy will have a 5-week venetoclax dose ramp-up period to reach the target dose of 400 mg QD. Following the venetoclax ramp-up period, Participants will receive 6 cycles of rituximab consisting of a single infusion on the first day of each 28-day cycle. Participants will continue to take their daily dose of venetoclax during the rituximab cycles. Participants who have not progressed following the completion of the 6 cycles will continue to receive venetoclax monotherapy until disease progression or for a maximum of 2 years from Cycle 1 Re-Treatment Day 1 of the Substudy.
  Interventions: Drug: Venetoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Bendamustine will be administered at a dose of 70 mg/m^2 via IV infusion on Days 1 and 2 of each 28-day cycle, for 6 cycles.
  Arms: Bendamustine + Rituximab
Drug: Venetoclax — Venetoclax will be administered at an initial dose of 20 mg via tablet orally QD, incremented weekly up to a maximum dose of 400 mg during a 5-week ramp-up period. Venetoclax will be continued at 400 mg QD from Week 6 (Day 1 of Cycle 1 of combination therapy) onwards up to disease progression (PD) or 2 years, whichever occurs first.
  R/C Substudy: venetoclax will be administered for 5-week dose ramp-up period to reach the target dose of 400 mg QD. Venetoclax will continue to be administered during the rituximab cycles until disease progression or for a maximum of 2 years from Cycle 1R/C Day 1 of the R/C Substudy.
  Other Names: GDC-0199, ABT-199
  Arms: Bendamustine + Rituximab Crossover Substudy; Venetoclax + Rituximab; Venetoclax + Rituximab Re-Treatment
Drug: Rituximab — Rituximab will be administered at a dose of 375 mg/m^2 via IV infusion on Day 1 of Cycle 1 and at a dose of 500 mg/m^2 on Day 1 of Cycles 2-6.
  R/C Substudy: Following the venetoclax ramp-up period, rituximab will be administered for 6 cycles consisting of a single infusion on the first day of each 28-day cycle.

SUMMARY:
The purpose of this open-label, multicenter, randomized, Phase III study is to evaluate the benefit of venetoclax in combination with rituximab compared with bendamustine in combination with rituximab in participants with relapsed or refractory CLL. Participants will be randomly assigned in 1:1 ratio to receive either venetoclax + rituximab (Arm A) or bendamustine + rituximab (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL per diagnostic criteria for relapsed or refractory CLL per the international workshop on chronic lymphocytic leukemia (iwCLL) guidelines
* Previously treated with 1-3 lines of therapy (example: completed greater than or equal to [>/=] 2 treatment cycles per therapy), including at least one standard chemotherapy-containing regimen
* Participants previously treated with bendamustine only if their duration of response was >/= 24 months
* Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to (</=) 1
* Adequate bone marrow function
* Adequate renal and hepatic function
* Participants must use effective birth control throughout study until at least 30 days after study treatment or 1 year after rituximab treatment, whichever is later; female participants must not be pregnant or breast-feeding
* For participants with the 17p deletion, previously treated with 1-3 lines of therapy, including at least one prior standard chemotherapy-containing regimen or at least one prior alemtuzumab-containing therapy

Inclusion Criteria R/C Substudy:

* Participants randomized to Arm A or Arm B with a confirmed disease progression of CLL per iwCLL criteria
* Participants who have not received new anti-CLL therapy following disease progression in Arm A or Arm B
* Adequate renal and hepatic function per laboratory reference range

Exclusion Criteria:

* Transformation of CLL to aggressive non-Hodgkin lymphoma or central nervous system (CNS) involvement by CLL
* Undergone an allogenic stem cell transplant
* A history of significant renal, neurologic, psychiatric, endocrine, metabolic, immunologic, cardiovascular or hepatic disease
* Hepatitis B or C or known human immunodeficiency virus (HIV) positive
* Receiving warfarin treatment
* Received an anti-CLL monoclonal antibody within 8 weeks prior to the first dose of study drug
* Received any anti-cancer or investigational therapy within 28 days prior to the first dose of study drug or has not recovered to less than Grade 2 clinically significant adverse effect(s)/toxicity(ies) of any previous therapy
* Received cytochrome P450 3A4 (CYP3A4) inhibitors (such as fluconazole, ketoconazole and clarithromycin) or inducers (such as rifampin, carbamazapine, phenytoin, St. John's Wort) within 7 days prior to the first dose of venetoclax
* History of prior venetoclax treatment
* Participants with another cancer, history of another cancer considered uncured on in complete remission for <5 years, or currently under treatment for another suspected cancer except non-melanoma skin cancer or carcinoma in situ of the cervix that has been treated or excised and is considered resolved
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Other clinically significant uncontrolled condition(s) including, but not limited to, systemic infection (viral, bacterial or fungal)
* Vaccination with a live vaccine within 28 days prior to randomization
* Consumed grapefruit or grapefruit products, seville oranges (including marmalade containing seville oranges), or star fruit within 3 days prior to the first dose of study treatment
* A cardiovascular disability status of New York Heart Association Class >/=3. Class 3 is defined as cardiac disease in which participants are comfortable at rest but have marked limitation of physical activity due to fatigue, palpitations, dyspnea, or anginal pain
* Major surgery within 30 days prior to the first dose of study treatment
* A participant who is pregnant or breastfeeding
* Known allergy to both xanthine oxidase inhibitors and rasburicase

Exclusion Criteria R/C Substudy:

* Transformation of CLL to aggressive NHL (e.g., Richter's transformation, prolymphocytic leukemia, or DLBCL) or CNS involvement by CLL
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, or fungal)
* Development of other malignancy since enrollment into the study, with the exception of curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia
* History of severe (i.e., requiring permanent discontinuation of prior rituximab therapy) prior allergic or anaphylactic reactions to rituximab
* Known HIV positivity
* Positive test results for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HbsAg] serology)
* Positive test results for hepatitis C virus (HCV; HCV antibody serology testing)
* Requires the use of warfarin (due to potential drug interactions that may potentially increase the exposure of warfarin)
* Has not recovered to less than Grade 2 clinically significant adverse effect(s)/toxicity(ies) of any previous therapy
* Received potent CYP3A4 inhibitors (such as fluconazole, ketoconazole, and clarithromycin) within 7 days prior to the first dose of study treatment
* Received potent CYP3A4 inducers (such as rifampin, carbamazepine, phenytoin, St. John's wort) within 7 days prior to the first dose of study treatment
* Consumed grapefruit or grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of study treatment
* A cardiovascular disability status of New York Heart Association Class >/= 3
* A significant history of renal, neurologic, psychiatric, endocrine, metabolic, immunologic, cardiovascular, or hepatic disease that, in the opinion of the investigator, would adversely affect the participants's participation in this study or interpretation of study outcomes
* Major surgery within 30 days prior to the first dose of study treatment
* A participant who is pregnant or breastfeeding
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Known allergy to both xanthine oxidase inhibitors and rasburicase
* Vaccination with a live vaccine within 28 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (111):
- United States (5):
  - University of California San Diego Medical Center, La Jolla, California
  - Henry Ford Health System, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center; Clinical Trials Office, New York, New York
  - Perlmutter Cancer Center NYU Langone Health, New York, New York
  - Huntsman Cancer Institute; University of Utah, Salt Lake City, Utah
- Australia (13):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Frankston Hospital, Frankston, Victoria
  - Monash Medical Centre; Haematology, Melbourne, Victoria
  - Slade Health Pharmacy, Mount Waverley, Victoria
  - Peter MacCallum Cancer Center, North Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - The Perth Blood Institute, Nedlands, Western Australia
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
  - Klinik Ottakring, Vienna
- Belgium (6):
  - ZNA Antwerpen; Department Hematology, Antwerp
  - Cliniques Universitaires Saint-Luc; Hematology, Brussels
  - AZ Groeninge, Kortrijk
  - UZ Leuven; Department Hematology, Leuven
  - CHU UCL Mont-Godinne, Mont-godinne
  - AZ Delta (Campus Rumbeke), Roeselare
- Canada (4):
  - Foothills Medical Centre; Centre Dept of Medical Clinical Neuroscience, Calgary, Alberta
  - Juravinski Cancer Clinic, Hamilton, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Saskatoon City Hospital;Saskatchewan Cancer Centre, Saskatoon, Saskatchewan
- Czechia (6):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultní nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- Denmark (5):
  - Herlev Hospital, Herlev
  - Rigshospitalet, København Ø
  - Odense Universitetshospital, Odense C
  - Sjællands Universitetshospital, Roskilde, Roskilde
  - Sygehus Lillebælt, Vejle, Vejle
- France (13):
  - Hôpital Morvan, Brest
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Hopital Claude Huriez - CHU Lille, Lille
  - Hopital Saint Eloi, Montpellier
  - CHU Nantes - Hôtel Dieu; Service Assistance Medicale à la Procreation, Nantes
  - Hopital Robert Debre, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers - Hopital La Miletrie, Poitiers
  - CHU de Rennes - Hopital de Pontchaillo, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Universitaire du Cancer - Oncopole Toulouse (IUCT-O), Toulouse
  - CHU Tours - Hôpital Bretonneau, Tours
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (3):
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Tübingen, Tübingen
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Központ; B?rgyógyászati Klinika, Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Pécs
  - Szegedi Tud.Egyetem Szent-Gyorgyi Albert Klin.Kozp., Szeged
- Italy (9):
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino; Radiology, Torino, Abruzzo
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico Bari, Bari, Apulia
  - Azienda Ospedaliero Universitaria San Martino, Genoa, Liguria
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo, Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; SC Farmacia Ospedale, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette Di Ancona, The Marches
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera Di Padova, Padua, Veneto
- Netherlands (7):
  - Amsterdam UMC, Locatie VUMC; Neurology, Amsterdam
  - Amsterdam UMC Location AMC, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordwijk; Internal Medicine, Hemato-Oncology, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - Leids Universitair Medisch Centrum; Cardiology, Leiden
  - Erasmus Medisch Centrum, Rotterdam
  - UMC Utrecht, Utrecht
- New Zealand (4):
  - North Shore Hospital; Haematolgy, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital NZ, Christchurch
  - Baxter Healthcare, Mount Wellington
- Poland (6):
  - SP ZOZ Zespol Szpitali Miejskich w Chorzowie, Chorzów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Szpital Wojewodzki w Opolu, Opole
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Zabrze
- Russia (5):
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow, Moscow Oblast
  - SRI of Hematology and Transfusiology, Saint Petersburg, Sankt-Peterburg
  - North-West Federal Medical Research Center n.a. V.A. Almazov, Saint Petersburg, Sankt-Peterburg
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary?s Hospital, Seoul
- Spain (5):
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona; Hematology, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
- Sweden (2):
  - Skånes Universitetssjukhus, Lund
  - Akademiska Sjukhuset, Uppsala
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (4):
  - Bristol Haematology and Oncology centre, Bristol
  - The Christie, Manchester
  - Southampton General Hospital, Southampton
  - Singleton Hospital; Pharmacy Department, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Kater AP, Harrup R, Kipps TJ, Eichhorst B, Owen CJ, Assouline S, Lamanna N, Robak T, de la Serna J, Jaeger U, Cartron G, Montillo M, Mellink C, Langerak AW, Chyla B, Popovic R, Jiang Y, Millen R, Lefebure M, Thadani-Mulero M, Boyer M, Seymour JF. The MURANO study: final analysis and retreatment/crossover substudy results of VenR for patients with relapsed/refractory CLL. Blood. 2025 Jun 5;145(23):2733-2745. doi: 10.1182/blood.2024025525. PMID 40009494
- [Derived] Badawi M, Chen X, Marroum P, Suleiman AA, Mensing S, Koenigsdorfer A, Schiele JT, Palenski T, Samineni D, Hoffman D, Menon R, Salem AH. Bioavailability Evaluation of Venetoclax Lower-Strength Tablets and Oral Powder Formulations to Establish Interchangeability with the 100 mg Tablet. Clin Drug Investig. 2022 Aug;42(8):657-668. doi: 10.1007/s40261-022-01172-4. Epub 2022 Jul 13. PMID 35829925
- [Derived] Seymour JF, Kipps TJ, Eichhorst BF, D'Rozario J, Owen CJ, Assouline S, Lamanna N, Robak T, de la Serna J, Jaeger U, Cartron G, Montillo M, Mellink C, Chyla B, Panchal A, Lu T, Wu JQ, Jiang Y, Lefebure M, Boyer M, Kater AP. Enduring undetectable MRD and updated outcomes in relapsed/refractory CLL after fixed-duration venetoclax-rituximab. Blood. 2022 Aug 25;140(8):839-850. doi: 10.1182/blood.2021015014. PMID 35605176
- [Derived] Kater AP, Wu JQ, Kipps T, Eichhorst B, Hillmen P, D'Rozario J, Assouline S, Owen C, Robak T, de la Serna J, Jaeger U, Cartron G, Montillo M, Dubois J, Eldering E, Mellink C, Van Der Kevie-Kersemaekers AM, Kim SY, Chyla B, Punnoose E, Bolen CR, Assaf ZJ, Jiang Y, Wang J, Lefebure M, Boyer M, Humphrey K, Seymour JF. Venetoclax Plus Rituximab in Relapsed Chronic Lymphocytic Leukemia: 4-Year Results and Evaluation of Impact of Genomic Complexity and Gene Mutations From the MURANO Phase III Study. J Clin Oncol. 2020 Dec 1;38(34):4042-4054. doi: 10.1200/JCO.20.00948. Epub 2020 Sep 28. PMID 32986498
- [Derived] Kater AP, Seymour JF, Hillmen P, Eichhorst B, Langerak AW, Owen C, Verdugo M, Wu J, Punnoose EA, Jiang Y, Wang J, Boyer M, Humphrey K, Mobasher M, Kipps TJ. Fixed Duration of Venetoclax-Rituximab in Relapsed/Refractory Chronic Lymphocytic Leukemia Eradicates Minimal Residual Disease and Prolongs Survival: Post-Treatment Follow-Up of the MURANO Phase III Study. J Clin Oncol. 2019 Feb 1;37(4):269-277. doi: 10.1200/JCO.18.01580. Epub 2018 Dec 3. PMID 30523712
- [Derived] Seymour JF, Kipps TJ, Eichhorst B, Hillmen P, D'Rozario J, Assouline S, Owen C, Gerecitano J, Robak T, De la Serna J, Jaeger U, Cartron G, Montillo M, Humerickhouse R, Punnoose EA, Li Y, Boyer M, Humphrey K, Mobasher M, Kater AP. Venetoclax-Rituximab in Relapsed or Refractory Chronic Lymphocytic Leukemia. N Engl J Med. 2018 Mar 22;378(12):1107-1120. doi: 10.1056/NEJMoa1713976. PMID 29562156
- [Derived] Jones AK, Freise KJ, Agarwal SK, Humerickhouse RA, Wong SL, Salem AH. Clinical Predictors of Venetoclax Pharmacokinetics in Chronic Lymphocytic Leukemia and Non-Hodgkin's Lymphoma Patients: a Pooled Population Pharmacokinetic Analysis. AAPS J. 2016 Sep;18(5):1192-1202. doi: 10.1208/s12248-016-9927-9. Epub 2016 May 27. PMID 27233802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 389 participants took part in the study across 109 investigative sites in 20 countries i.e., Korea, Taiwan, Australia, New Zealand, Czech Republic, Hungary, Poland, Russia, Canada, United States of America, Austria, Belgium, Germany, Denmark, Spain, France, United Kingdom, Italy, Netherlands and Sweden from 17 March 2014 to 03 August 2022. The trial consisted of a main study and an optional Retreatment/Crossover (R/C) sub study.
Pre-assignment Details: Of the 389 participants enrolled 7 participants in the bendamustine + rituximab (BR) arm did not receive a valid dose of study treatment.
Groups:
- Bendamustine + Rituximab Main Study: Participants received bendamustine at a dose of 70 milligrams per meter square (mg/m^2) via intravenous (IV) infusion on Days 1 and 2 of each 28-day cycle for 6 cycles, in combination with rituximab at a dose of 375 mg/m^2 via IV infusion on Day 1 of Cycle 1 and at a dose of 500 mg/m^2 on Day 1 of Cycles 2-6.
- Venetoclax + Rituximab Main Study: Participants were initially placed on a venetoclax ramp-up period of 5 weeks and received an initial dose of 20 mg via tablet orally once daily (QD) for initial 1 to 7 days, then venetoclax dose was incremented weekly up to a maximum dose of 400 mg, orally, QD. Participants continued receiving venetoclax at a dose of 400 mg, orally, QD from Week 6 (Day 1 of Cycle 1 of combination therapy) onwards up to progressive disease (PD) or 2 years, whichever occurred first, as directed by the investigator, in combination with rituximab at a dose of 375 mg/m^2 via IV infusion on Day 1 of Cycle 1 and at a dose of 500 mg/m^2 on Day 1 of Cycles 2-6.
- Bendamustine + Rituximab Crossover Substudy: Participants who entered the crossover substudy had a 5-week venetoclax dose ramp-up period to reach the target dose of 400 mg QD. Following the venetoclax ramp-up period, participants received 6 cycles of rituximab, 375 mg/m^2, as IV infusion on the Day 1 of each 28-day cycle. Participants who did not progress following the completion of the 6 cycles continued to receive venetoclax monotherapy until disease progression or for a maximum of 2 years from Cycle 1 crossover Day 1 of the substudy.
- Venetoclax + Rituximab Re-Treatment Substudy: Participants who entered the re-treatment substudy had a 5-week venetoclax dose ramp-up period to reach the target dose of 400 mg QD. Following the venetoclax ramp-up period, participants received 6 cycles of rituximab consisting of a single infusion on the first day of each 28-day cycle. Participants who did not progress following the completion of the 6 cycles continued to receive venetoclax monotherapy until disease progression or for a maximum of 2 year from Cycle 1 re-treatment Day 1 of the substudy.
Period: Main Study
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study | Bendamustine + Rituximab Crossover Substudy | Venetoclax + Rituximab Re-Treatment Substudy
Started | 195 | 194 | 0 | 0
Safety Evaluable (SE) Population (SE population included all randomized participants who received at least one dose of study treatment with participants grouped according to the actual treatment received.) | 188 | 194 | 0 | 0
Completed | 71 | 118 | 0 | 0
Not Completed | 124 | 76 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 83 | 52 | 0 | 0
Not completed — Lost to Follow-up | 4 | 5 | 0 | 0
Not completed — Physician Decision | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 26 | 11 | 0 | 0
Not completed — Reason not Specified | 0 | 6 | 0 | 0
Not completed — Randomized but not Dosed | 8 | 0 | 0 | 0
Period: Re-Treatment/Crossover (R/C) Substudy
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study | Bendamustine + Rituximab Crossover Substudy | Venetoclax + Rituximab Re-Treatment Substudy
Started | 0 (Following the end of main study, participants who had progressed clinically and were in need of therapy participated in the Re-Treatment/Crossover Substudy at the discretion of the investigator.) | 0 (Following the end of main study, participants who had progressed clinically and were in need of therapy participated in the Re-Treatment/Crossover Substudy at the discretion of the investigator.) | 9 (9 participants from BR arm entered R/C substudy.) | 25 (25 participants from VR arm entered R/C substudy.)
Completed | 0 | 0 | 7 | 15
Not Completed | 0 | 0 | 2 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants, with participants grouped according to randomized treatment group, regardless of the actual treatment received.
Groups:
- Venetoclax + Rituximab Main Study: Participants were initially placed on a venetoclax ramp-up period of 5 weeks and received an initial dose of 20 mg via tablet orally once daily (QD) for initial 1 to 7 days, then venetoclax dose was incremented weekly up to a maximum dose of 400 mg, orally, QD. Participants continued receiving venetoclax at a dose of 400 mg, orally, QD from Week 6 (Day 1 of Cycle 1 of combination therapy) onwards up to PD or 2 years, whichever occurred first, as directed by the investigator, in combination with rituximab at a dose of 375 mg/m^2 via IV infusion on Day 1 of Cycle 1 and at a dose of 500 mg/m^2 on Day 1 of Cycles 2-6.
- Total: Total of all reporting groups
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study | Total
Number analyzed (Participants) | 195 | 194 | 389
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (9.6) | 63.9 (10.5) | 64.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 58 | 102
  Male | 151 | 136 | 287
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 186 | 186 | 372
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 178 | 181 | 359
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With PD as Assessed by the Investigator Using Standard International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Guidelines or Death
Description: Assessment of response was performed by the investigator according to the iwCLL guidelines. PD was defined as occurrence of one of the following events: appearance of any new extra nodal lesion; new palpable lymph node (greater than [>] 1.5 centimeters [cm]); unequivocal progression of non-target lesion; an increase of greater than or equal to (>/=) 50 percent (%) compared to baseline in splenomegaly, hepatomegaly, number of blood lymphocytes with lymphocyte count >/=5000 per microliter (mcL), or in longest diameter of any extra nodal lesion; transformation to a more aggressive histology; decrease of >/=50% compared to baseline in platelet or neutrophil count; or decrease in hemoglobin level by >2 grams per deciliter (g/dL) or to less than [<] 10 g/dL. Percentages are rounded off.
Time Frame: Baseline up to PD or death from any cause, whichever occurred first (up to approximately 8 years 5 months)
Population: ITT population included all randomized participants, with participants grouped according to randomized treatment group, regardless of the actual treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants | 88.7 | 70.1

2. Primary Outcome: Progression-Free Survival (PFS) as Assessed by the Investigator Using Standard iwCLL Guidelines
Description: PFS was defined as the time from randomization until first occurrence of PD/relapse as assessed by the investigator using iwCLL guidelines, or death from any cause, whichever occurred first. PD: occurrence of one of the following: new lesion; new palpable lymph node (>1.5 cm); unequivocal progression of non-target lesion; increase of >/=50% in splenomegaly, hepatomegaly, blood lymphocytes with count >/=5000/mcL, longest diameter of any lesion; transformation to more aggressive histology; decrease of >/=50% in platelet or neutrophil count, or hemoglobin level by >2 g/dL or to <10 g/dL. Participants who had not progressed, relapsed, or died at the time of analysis, were censored on the date of last assessment. In case of no disease assessment after baseline, PFS was censored at the time of randomization+1 day. The median PFS was estimated using Kaplan-Meier method and the 95% confidence interval (CI) was computed using method of Brookmeyer and Crowley.
Time Frame: Baseline up to PD or death, whichever occurred first (up to approximately 8 years 5 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
months | 17.0 [15.5 to 21.7] | 54.7 [52.3 to 59.9]
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Stratified analysis: 17p deletion, risk status, geographic region; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.18 to 0.29] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Unstratified Analysis; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.25, 95% CI 2-sided [0.19 to 0.31] — Hazard ratio was estimated by Cox regression model

3. Secondary Outcome: Percentage of Participants With PD or Death as Assessed by the Independent Review Committee (IRC) Using Standard iwCLL Guidelines
Description: Assessment of response was performed by the IRC according to the iwCLL guidelines. PD was defined as occurrence of one of the following events: appearance of any new extra nodal lesion; new palpable lymph node (>1.5 cm); unequivocal progression of non-target lesion; an increase of >/=50% compared to baseline in splenomegaly, hepatomegaly, number of blood lymphocytes with lymphocyte count >/=5000/mcL, or in longest diameter of any extra nodal lesion; transformation to a more aggressive histology; decrease of >/=50% compared to baseline in platelet or neutrophil count; or decrease in hemoglobin level by >2 g/dL or to <10 g/dL. No new IRC data was generated post the primary analysis.
Time Frame: Baseline up to PD or death, whichever occurred first (up to approximately 3 years)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants | 54.4 | 18.0

4. Secondary Outcome: PFS as Assessed by the IRC Using Standard iwCLL Guidelines
Description: PFS was defined as the time from randomization until first occurrence of PD/relapse as assessed by the IRC using iwCLL guidelines, or death from any cause, whichever occurred first. PD: occurrence of one of the following: new lesion; new palpable lymph node (>1.5 cm); unequivocal progression of non-target lesion; increase of >/=50% in splenomegaly, hepatomegaly, blood lymphocytes with count >/=5000/mcL, longest diameter of any lesion; transformation to more aggressive histology; decrease of >/=50% in platelet or neutrophil count, or hemoglobin level by >2 g/dL or to <10 g/dL. Participants who had not progressed, relapsed, or died at the time of analysis, were censored on the date of last assessment. In case of no disease assessment after baseline, PFS was censored at the time of randomization+1 day. The median PFS was estimated using Kaplan-Meier method and the 95% CI was computed using method of Brookmeyer and Crowley. No new IRC data was generated post the primary analysis.
Time Frame: Baseline up to PD or death, whichever occurred first (up to approximately 3 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
months | 18.1 [15.8 to 22.3] | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to low number of participants with an event.
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Stratified Analysis; Stratification factors: 17p deletion, risk status, geographic region; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.19, 95% CI 2-sided [0.13 to 0.28] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Unstratified Analysis; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.20, 95% CI 2-sided [0.14 to 0.30] — Hazard ratio was estimated by Cox regression model

5. Secondary Outcome: Percentage of Participants With PD or Death as Assessed by the Investigator Using Standard iwCLL Guidelines in Participants With 17p Deletion as Identified by Fluorescence In-situ Hybridization (FISH) Test
Description: Assessment of response was performed by the investigator according to the iwCLL guidelines. PD was defined as occurrence of one of the following events: appearance of any new extra nodal lesion; new palpable lymph node (>1.5 cm); unequivocal progression of non-target lesion; an increase of >/=50% compared to baseline in splenomegaly, hepatomegaly, number of blood lymphocytes with lymphocyte count >/=5000/mcL, or in longest diameter of any extra nodal lesion; transformation to a more aggressive histology; decrease of >/=50% compared to baseline in platelet or neutrophil count; or decrease in hemoglobin level by >2 g/dL or to <10 g/dL. Percentages are rounded off.
Time Frame: Baseline up to PD or death, whichever occurred first (up to approximately 8 years 5 months)
Population: Analysis was performed on ITT population participants with 17p deletion as identified by FISH test.
Measure: Number; unit: percentage of participants
Groups:
- Bendamustine + Rituximab 17p Del. Population: Participants received bendamustine at a dose of 70 mg/m^2 via IV infusion on Days 1 and 2 of each 28-day cycle for 6 cycles, in combination with rituximab at a dose of 375 mg/m^2 via IV infusion on Day 1 of Cycle 1 and at a dose of 500 mg/m^2 on Day 1 of Cycles 2-6. Only participants with 17p deletion as identified by FISH test were included.
- Venetoclax + Rituximab 17p Del. Population: Participants were initially placed on a venetoclax ramp-up period of 4 to 5 weeks, and received an initial dose of 20 mg via tablet orally QD for initial 1 to 7 days, then venetoclax dose was incremented weekly up to a maximum dose of 400 mg via tablet orally QD. Participants continued receiving venetoclax at a dose of 400 mg via tablet orally QD from Week 6 (Day 1 of Cycle 1 of combination therapy) onwards up to PD or 2 years, whichever occurred first, as directed by the investigator, in combination with rituximab at a dose of 375 mg/m^2 via IV infusion on Day 1 of Cycle 1 and at a dose of 500 mg/m^2 on Day 1 of Cycles 2-6. Only participants with 17p deletion as identified by FISH test were included.
Arm/Group | Bendamustine + Rituximab 17p Del. Population | Venetoclax + Rituximab 17p Del. Population
Number analyzed (Participants) | 46 | 46
percentage of participants | 80.4 | 80.4

6. Secondary Outcome: PFS as Assessed by the Investigator Using Standard iwCLL Guidelines in Participants With 17p Deletion as Identified by FISH Test
Description: PFS was defined as the time from randomization until first occurrence of PD/relapse as assessed by the investigator using iwCLL guidelines, or death from any cause, whichever occurred first. PD: occurrence of one of the following: new lesion; new palpable lymph node (>1.5 cm); unequivocal progression of non-target lesion; increase of >/=50% in splenomegaly, hepatomegaly, blood lymphocytes with count >/=5000/mcL, longest diameter of any lesion; transformation to more aggressive histology; decrease of >/=50% in platelet or neutrophil count, or hemoglobin level by >2 g/dL or to <10 g/dL. Participants who had not progressed, relapsed, or died at the time of analysis, were censored on the date of last assessment. In case of no disease assessment after baseline, PFS was censored at the time of randomization+1 day. The median PFS was estimated using Kaplan-Meier method and the 95% CI was computed using method of Brookmeyer and Crowley.
Time Frame: Baseline up to PD or death, whichever occurred first (up to approximately 8 years 5 months)
Population: Analysis was performed on ITT population participants with 17p deletion as identified by FISH test.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine + Rituximab 17p Del. Population | Venetoclax + Rituximab 17p Del. Population
Number analyzed (Participants) | 46 | 46
months | 15.4 [10.0 to 21.0] | 47.9 [37.4 to 59.9]
Statistical Analysis 1: Comparison: Bendamustine + Rituximab 17p Del. Population vs Venetoclax + Rituximab 17p Del. Population; Stratified Analysis; Stratification factor: geographic region; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.21 to 0.57] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Bendamustine + Rituximab 17p Del. Population vs Venetoclax + Rituximab 17p Del. Population; Unstratified Analysis; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.22 to 0.56] — Hazard ratio was estimated by Cox regression model

7. Secondary Outcome: Percentage of Participants With PD or Death as Assessed by the IRC Using Standard iwCLL Guidelines in Participants With 17p Deletion as Identified by FISH Test
Description: as for outcome 3
Time Frame: Baseline up to PD or death, whichever occurred first (up to approximately 3 years)
Population: Analysis was performed on ITT population participants with 17p deletion as identified by FISH test.
Measure: Number; unit: percentage of participants
Arm/Group | Bendamustine + Rituximab 17p Del. Population | Venetoclax + Rituximab 17p Del. Population
Number analyzed (Participants) | 46 | 46
percentage of participants | 47.8 | 19.6

8. Secondary Outcome: PFS as Assessed by the IRC Using Standard iwCLL Guidelines in Participants With 17p Deletion as Identified by FISH Test
Description: as for outcome 4
Time Frame: Baseline up to PD or death, whichever occurred first (up to approximately 3 years)
Population: Analysis was performed on ITT population participants with 17p deletion as identified by FISH test.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine + Rituximab 17p Del. Population | Venetoclax + Rituximab 17p Del. Population
Number analyzed (Participants) | 46 | 46
months | 16.1 [13.6 to 22.3] | NA [27.6 to NA] — Median and Upper Limit of 95% CI could not be estimated due to low number of participants with an event.
Statistical Analysis 1: Comparison: Bendamustine + Rituximab 17p Del. Population vs Venetoclax + Rituximab 17p Del. Population; Stratified Analysis; Stratification factor: geographic region; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.09 to 0.49] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Bendamustine + Rituximab 17p Del. Population vs Venetoclax + Rituximab 17p Del. Population; Unstratified Analysis; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.09 to 0.46] — Hazard ratio was estimated by Cox regression model

9. Secondary Outcome: Percentage of Participants With Best Overall Response of Complete Response (CR), CR With Incomplete Bone Marrow Recovery (CRi), Nodular Partial Response (nPR), or Partial Response (PR) as Assessed by the Investigator Using iwCLL Guidelines
Description: Response was assessed by investigator according to iwCLL guidelines and was confirmed by repeat assessment >/=4 weeks after initial documentation. CR: peripheral blood lymphocytes <4000/mcL; absence of any new lesion, nodal disease, lymphadenopathy, hepatomegaly, splenomegaly, and constitutional symptoms; neutrophils >1500/mcL, platelets >100000/mcL, hemoglobin >11.0 g/dL without need for transfusion or exogenous growth factors; normocellular bone marrow with <30% lymphocytes; no lymphoid nodules. CRi: fulfilling all CR criteria but persistent cytopenia. PR: >/=50% reduction in two of following: peripheral blood lymphocytes, lymphadenopathy, spleen and/or liver enlargement; and 1 of following: neutrophils >1500/mcL, platelets >100000/mcL, hemoglobin >11.0 g/dL or >/=50% improvement without need for transfusion or exogenous growth factors. nPR: fulfilling all CR criteria but presence of lymphoid nodules. 95% CI was computed using Pearson-Clopper method.Percentages are rounded off.
Time Frame: Baseline up to approximately 8 years 5 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants
  CR | 8.2 [4.76 to 12.98] | 26.3 [20.24 to 33.07]
  CRi | 0.5 [0.01 to 2.82] | 1.5 [0.32 to 4.45]
  nPR | 6.2 [3.22 to 10.50] | 3.6 [1.46 to 7.29]
  PR | 52.8 [45.56 to 59.99] | 61.9 [54.62 to 68.72]
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Difference in Response Rates = 25.61, 95% CI 2-sided [17.88 to 33.33] — 95% CI for rates were constructed using Pearson- Clopper method. 95% CI for difference in rates were constructed using Anderson-Hauck method
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; Odds Ratio (OR) = 7.81, 95% CI 2-sided [3.97 to 15.37] — OR was estimated using logistic regression model. The 95% CI was computed using Wald test

10. Secondary Outcome: Percentage of Participants With Best Overall Response of CR, CRi, nPR, or PR as Assessed by the IRC Using iwCLL Guidelines
Description: Response was assessed by IRC according to iwCLL guidelines and was confirmed by repeat assessment >/=4 weeks after initial documentation. CR: peripheral blood lymphocytes <4000/mcL; absence of any new lesion, nodal disease, lymphadenopathy, hepatomegaly, splenomegaly, constitutional symptoms; neutrophils >1500/mcL, platelets >100000/mcL, hemoglobin >11.0 g/dL without need for transfusion or exogenous growth factors; normocellular bone marrow with <30% lymphocytes; no lymphoid nodules. CRi: fulfilling all CR criteria but persistent cytopenia. PR: >/=50% reduction in 2 of following: peripheral blood lymphocytes, lymphadenopathy, spleen and/or liver enlargement; 1 of following: neutrophils >1500/mcL, platelets >100000/mcL, hemoglobin >11.0 g/dL or >/=50% improvement without need for transfusion or exogenous growth factors. nPR: fulfilling all CR criteria but presence of lymphoid nodules. 95% CI was computed using Pearson-Clopper method.No new IRC data was generated post primary analysis.
Time Frame: Baseline up to last FUV (up to approximately 3 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants | 67.7 [60.64 to 74.20] | 93.3 [88.81 to 96.38]
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Difference in Response Rates = 25.61, 95% CI 2-sided [17.88 to 33.33] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; Odds Ratio (OR) = 7.81, 95% CI 2-sided [3.97 to 15.37] — OR was estimated using logistic regression model. The 95% CI was computed using Wald test

11. Secondary Outcome: Percentage of Participants With Overall Response of CR, Cri, nPR, or PR at End of Combination Treatment Visit as Assessed by the Investigator Using iwCLL Guidelines
Description: Response was assessed by investigator according to iwCLL guidelines and was confirmed by repeat assessment >/=4 weeks after initial documentation. CR: peripheral blood lymphocytes <4000/mcL; absence of any new lesion, nodal disease, lymphadenopathy, hepatomegaly, splenomegaly, and constitutional symptoms; neutrophils >1500/mcL, platelets >100000/mcL, hemoglobin >11.0 g/dL without need for transfusion or exogenous growth factors; normocellular bone marrow with <30% lymphocytes; no lymphoid nodules. CRi: fulfilling all CR criteria but persistent cytopenia. PR: >/=50% reduction in 2 of following: peripheral blood lymphocytes, lymphadenopathy, spleen and/or liver enlargement; and 1 of following: neutrophils >1500/mcL, platelets >100000/mcL, hemoglobin >11.0 g/dL or >/=50% improvement without need for transfusion or exogenous growth factors. nPR: fulfilling all CR criteria but presence of lymphoid nodules. 95% CI was computed using Pearson-Clopper method. Percentages are rounded off.
Time Frame: End of combination treatment response (EoCTR) visit (8 to 12 weeks after Cycle [C] 6 Day [1]); Cycle length = 28 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants | 63.1 [55.89 to 69.86] | 88.1 [82.74 to 92.33]
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Difference in Response Rates = 25.07, 95% CI 2-sided [16.63 to 33.51] — The 95% CI was computed using Anderson-Hauck method
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; Odds Ratio (OR) = 4.59, 95% CI 2-sided [2.68 to 7.88] — OR was estimated using logistic regression model. The 95% CI was computed using Wald test

12. Secondary Outcome: Percentage of Participants With Overall Response of CR, Cri, nPR, or PR at End of Combination Treatment Visit as Assessed by the IRC Using iwCLL Guidelines
Description: Response was assessed by the IRC according to the iwCLL guidelines and was confirmed by repeat assessment >/=4 weeks after initial documentation. CR: peripheral blood lymphocytes <4000/mcL; absence of any new lesion, nodal disease, lymphadenopathy, hepatomegaly, splenomegaly, and constitutional symptoms; neutrophils >1500/mcL, platelets >100000/mcL, hemoglobin >11.0 g/dL without need for transfusion or exogenous growth factors; normocellular bone marrow with <30% lymphocytes; no lymphoid nodules. CRi: fulfilling all CR criteria but persistent cytopenia. PR: >/=50% reduction in two of the following: peripheral blood lymphocytes, lymphadenopathy, spleen and/or liver enlargement; and one of the following: neutrophils >1500/mcL, platelets >100000/mcL, hemoglobin >11.0 g/dL or >/=50% improvement without need for transfusion or exogenous growth factors. nPR: fulfilling all CR criteria but presence of lymphoid nodules. The 95% CI was computed using Pearson-Clopper method.
Time Frame: EoCTR visit (8 to 12 weeks after C6D1); Cycle length = 28 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants | 62.6 [55.37 to 69.37] | 87.1 [81.57 to 91.48]
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Difference in Response Rates = 24.55, 95% CI 2-sided [16.00 to 33.10] — The 95% CI was computed using Anderson-Hauck method
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; Odds Ratio (OR) = 4.59, 95% CI 2-sided [2.68 to 7.85] — OR was estimated using logistic regression model. The 95% CI was computed using Wald test

13. Secondary Outcome: Percentage of Participants Who Died
Description: Percentage of participants who died from any cause, during the study, was reported. Percentage is rounded off.
Time Frame: Baseline up to approximately 8 years 5 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants | 43.1 | 30.9

14. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. Participants alive at the time of the analysis were censored at the date when they were last known to be alive as documented by the investigator. The median OS was estimated using Kaplan-Meier method and the 95% CI was computed using method of Brookmeyer and Crowley.
Time Frame: Baseline up to approximately 8 years 5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
months | 87.8 [70.1 to NA] — Upper limit was not estimable due to low number of participants with event. | NA [NA to NA] — Median, lower limit and upper limit were not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority — Stratified Analysis; Stratification factors: 17p deletion, risk status, geographic region; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.37 to 0.74] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Unstratified Analysis; Test type: Superiority; p = 0.0003, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.39 to 0.76] — Hazard ratio was estimated by Cox regression model

15. Secondary Outcome: Percentage of Participants With PD/Relapse, Start of a New Anti-Chronic Lymphocytic Leukemia (CLL) Therapy, or Death as Assessed by the Investigator Using iwCLL Guidelines
Description: Percentage of participants with PD/relapse, death from any cause, or start of a new non-protocol-specified anti-CLL therapy as assessed by the investigator, during the study, was reported. PD was defined as occurrence of one of the following events: appearance of any new extra nodal lesion; new palpable lymph node (>1.5 cm); unequivocal progression of non-target lesion; an increase of >/=50% compared to baseline in splenomegaly, hepatomegaly, number of blood lymphocytes with lymphocyte count >/=5000/mcL, or in longest diameter of any extra nodal lesion; transformation to a more aggressive histology; decrease of >/=50% compared to baseline in platelet or neutrophil count; or decrease in hemoglobin level by >2 g/dL or to <10 g/dL. Percentages are rounded off.
Time Frame: Baseline up to PD/relapse, start of a new anti-CLL therapy, or death from any cause, whichever occurred first (approximately 8 years 5 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants | 89.2 | 71.1

16. Secondary Outcome: Event-Free Survival (EFS) as Assessed by the Investigator Using iwCLL Guidelines
Description: EFS was defined as the time from date of randomization until the date of PD/relapse, start of a new non-protocol-specified anti-CLL therapy, or death from any cause, whichever occurred first, as assessed by the investigator. PD: occurrence of one of the following: new lesion; new palpable lymph node (>1.5 cm); unequivocal progression of non-target lesion; increase of >/=50% in splenomegaly, hepatomegaly, blood lymphocytes with count >/=5000/mcL, longest diameter of any lesion; transformation to more aggressive histology; decrease of >/=50% in platelet or neutrophil count, or hemoglobin level by >2 g/dL or to <10 g/dL. Participants without any of the specified event at the time of analysis were censored at the date of last adequate response assessment. In case of no post-baseline response assessment, participants were censored at the randomization date. The median EFS was estimated using Kaplan-Meier method and the 95% CI was computed using method of Brookmeyer and Crowley.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
months | 16.4 [14.2 to 21.0] | 53.7 [48.5 to 59.3]
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Stratified Analysis; Stratification factors: 17p deletion, risk status, geographic region; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.22, 95% CI 2-sided [0.17 to 0.29] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Unstratified Analysis; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.25, 95% CI 2-sided [0.19 to 0.31] — Hazard ratio was estimated by Cox regression model

17. Secondary Outcome: Percentage of Participants With PD or Death Among Participants With Best Overall Response of CR, CRi, nPR, or PR as Assessed by the Investigator Using iwCLL Guidelines
Description: Percentage of participants with PD as assessed by the investigator according to the iwCLL guidelines or death from any cause during the study was reported. PD was defined as occurrence of one of the following events: appearance of any new extra nodal lesion; new palpable lymph node (>1.5 cm); unequivocal progression of non-target lesion; an increase of >/=50% compared to baseline in splenomegaly, hepatomegaly, number of blood lymphocytes with lymphocyte count >/=5000/mcL, or in longest diameter of any extra nodal lesion; transformation to a more aggressive histology; decrease of >/=50% compared to baseline in platelet or neutrophil count; or decrease in hemoglobin level by >2 g/dL or to <10 g/dL. CR, CRi, nPR, and PR have been defined in previous outcomes, and are not repeated here due to space constraint. Percentage is rounded off.
Time Frame: From time of achieving best overall response until PD or death from any cause, whichever occurred first (up to approximately 8 years 5 months)
Population: Analysis was performed on ITT population participants who had best overall response of CR, CRi, nPR, or PR.
Measure: Number; unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 132 | 181
percentage of participants | 95.5 | 68.5

18. Secondary Outcome: Duration of Responses (DOR) as Assessed by the Investigator Using iwCLL Guidelines
Description: DOR was defined as the time from first occurrence of a documented response of CR, CRi, nPR, or PR until PD/relapse, as assessed by the investigator according to the iwCLL guidelines, or death from any cause. PD: occurrence of one of the following: new lesion; new palpable lymph node (>1.5 cm); unequivocal progression of non-target lesion; increase of >/=50% in splenomegaly, hepatomegaly, blood lymphocytes with count >/=5000/mcL, longest diameter of any lesion; transformation to more aggressive histology; decrease of >/=50% in platelet or neutrophil count, or hemoglobin level by >2 g/dL or to <10 g/dL. Participants without PD or death after response were censored at the last date of adequate response assessment. The median DOR was estimated using Kaplan-Meier method and the 95% CI was computed using method of Brookmeyer and Crowley. CR, CRi, nPR, and PR have been defined in previous outcomes, and are not repeated here due to space constraint.
Time Frame: as for outcome 17
Population: Analysis was performed on ITT population participants who had best overall response of CR, CRi, nPR, or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 132 | 181
months | 19.1 [16.1 to 23.6] | 53.6 [49.1 to 57.0]

19. Secondary Outcome: Percentage of Participants With Start of New Anti-CLL Treatment or Death as Assessed by the Investigator
Description: Percentage of participants with start of new non-protocol-specified anti-CLL therapy, as assessed by the investigator, or death from any cause, during the study, was reported. Percentage is rounded off.
Time Frame: Baseline up to start of new ani-CLL therapy or death, whichever occurred first (up to approximately 8 years 5 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants | 81.5 | 62.4

20. Secondary Outcome: Time to New Anti-CLL Treatment (TTNT) as Assessed by the Investigator
Description: TTNT was defined as the time from randomization until start of new non-protocol-specified anti-CLL treatment or death from any cause. Participants without the event at the time of analysis were censored at the last visit date for this outcome measure analysis. The median TTNT was estimated using Kaplan-Meier method and the 95% CI was computed using method of Brookmeyer and Crowley.
Time Frame: Baseline up to start of new ani-CLL therapy or death, whichever occurred first (up to approximately 8 years 5 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
months | 24.0 [20.7 to 29.5] | 63.0 [56.1 to 73.6]
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Stratified Analysis; Stratification factors: 17p deletion, risk status, geographic region; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.23 to 0.39] — Hazard ratio was estimated by Cox regression model
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Unstratified Analysis; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.25 to 0.41] — Hazard ratio was estimated by Cox regression model

21. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Negativity in Peripheral Blood
Description: MRD-negativity was defined as the presence of <1 malignant B-cell per 10000 normal B-cells in a sample of at least 200000 B-cells, as assessed by the allele specific oligonucleotide polymerase chain reaction (ASO-PCR) and/or flow cytometry technique. Percentage of participants with MRD-negativity was reported. The 95% CI was computed using Pearson-Clopper method. Percentage is rounded off.
Time Frame: EoCTR visit (8 to 12 weeks after C6D1); Cycle length = 28 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants | 13.3 [8.90 to 18.92] | 62.4 [55.15 to 69.21]
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; p < .0001, Chi-squared; Difference in MRD Negativity Rates = 49.04, 95% CI 2-sided [40.44 to 57.64] — The 95% CI was computed using Anderson-Hauck method
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; Odds Ratio (OR) = 10.77, 95% CI 2-sided [6.50 to 17.85] — OR was estimated using logistic regression model. The 95% CI was computed using Wald test

22. Secondary Outcome: Percentage of Participants With MRD Negativity in Bone Marrow
Description: MRD-negativity was defined as the presence of <1 malignant B-cell per 10000 normal B-cells in a sample of at least 200000 B-cells, as assessed flow cytometry technique. Percentage of participants with MRD-negativity was reported. The 95% CI was computed using Pearson-Clopper method. Percentages are rounded off.
Time Frame: EoCTR visit (8 to 12 weeks after C6D1); Cycle length = 28 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 195 | 194
percentage of participants | 1.0 [0.12 to 3.66] | 14.4 [9.81 to 20.18]
Statistical Analysis 1: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; p < .0001, Chi-squared; Difference in MRD negative rates = 13.41, 95% CI 2-sided [7.99 to 18.82] — The 95% CI was computed using Anderson-Hauck method
Statistical Analysis 2: Comparison: Bendamustine + Rituximab Main Study vs Venetoclax + Rituximab Main Study; Test type: Superiority; Odds Ratio (OR) = 16.28, 95% CI 2-sided [3.82 to 69.35] — OR was estimated using logistic regression model. The 95% CI was computed using Wald test

23. Secondary Outcome: Plasma Venetoclax Concentrations
Time Frame: Pre-dose (0 hour, anytime before venetoclax administration) and 4 hours post-dose on D1 of Cycles 1 and 4; Cycle length = 28 days
Population: Pharmacokinetic (PK) evaluable population included all participants in the 'Venetoclax + Rituximab' arm who received at least one dose of venetoclax with at least one post-dose PK concentration result available. Here 'Number Analyzed' signifies the number of participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 184
micrograms per milliliter (mcg/mL)
  C1D1, Pre-dose: number analyzed (Participants) | 151
  C1D1, Pre-dose | 0.626 (0.540)
  C1D1, 4 hours Post-Dose: number analyzed (Participants) | 159
  C1D1, 4 hours Post-Dose | 1.34 (0.881)
  C4D1, Pre-dose: number analyzed (Participants) | 112
  C4D1, Pre-dose | 0.681 (0.745)
  C4D1, 4 hours Post-Dose: number analyzed (Participants) | 121
  C4D1, 4 hours Post-Dose | 1.34 (0.905)

24. Secondary Outcome: Change From Baseline in Monroe Dunaway (MD) Anderson Symptom Inventory (MDASI) Core Symptom Severity, Module Symptom Severity, and Interference Scores
Description: MDASI is a 25-item validated questionnaire consisting of 2 parts. Part 1: 19-items divided into 2 scales, Core Symptom Severity (average of Questions 1 to 13; total 13 items: pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, remembering things, lack of appetite, drowsiness, dry mouth, sadness, vomiting, and numbness) and Module Symptom Severity (average of Questions 14 to 19; total 6 items: night sweats, fevers and chills, lymph node swelling, diarrhea, bruising easy or bleeding, and constipation). Part 2: 6-items to assess Interference (symptom distress) (average of Questions 20 to 25; total 6 items: general activity, walking, work, mood, relations with other people, and enjoyment of life). Each item was rated from 0 to 10, with lower scores indicating better outcome. Total score for Core Symptom Severity, Module Symptom Severity, and Interference are reported which range from 0 to 10, with lower scores indicating better health-related quality of life (HRQoL).
Time Frame: Baseline, Days 1, 8, and 15 of Cycles 1, 2, and 3; Cycle length = 28 days
Population: Patient reported outcomes (PRO) evaluable population included all participants with baseline and at least one post-baseline PRO assessment. Here, 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure and 'Number Analyzed' = participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 117 | 42
units on a scale
  Baseline; Mean core symptom severity: number analyzed (Participants) | 116 | 42
  Baseline; Mean core symptom severity | 1.76 (1.55) | 1.55 (1.31)
  Change at C1D1; Mean core symptom severity: number analyzed (Participants) | 116 | 36
  Change at C1D1; Mean core symptom severity | 0.00 (0.00) | -0.08 (0.98)
  Change at C1D8; Mean core symptom severity: number analyzed (Participants) | 107 | 36
  Change at C1D8; Mean core symptom severity | 0.26 (1.34) | -0.30 (0.84)
  Change at C1D15; Mean core symptom severity: number analyzed (Participants) | 104 | 33
  Change at C1D15; Mean core symptom severity | 0.00 (1.31) | -0.27 (0.93)
  Change at C2D1; Mean core symptom severity: number analyzed (Participants) | 101 | 35
  Change at C2D1; Mean core symptom severity | -0.23 (1.30) | -0.33 (0.91)
  Change at C2D8; Mean core symptom severity: number analyzed (Participants) | 91 | 36
  Change at C2D8; Mean core symptom severity | 0.17 (1.59) | -0.45 (0.91)
  Change at C2D15; Mean core symptom severity: number analyzed (Participants) | 90 | 37
  Change at C2D15; Mean core symptom severity | -0.13 (1.53) | -0.53 (0.90)
  Change at C3D1; Mean core symptom severity: number analyzed (Participants) | 89 | 36
  Change at C3D1; Mean core symptom severity | -0.26 (1.60) | -0.40 (1.13)
  Change at C3D8; Mean core symptom severity: number analyzed (Participants) | 72 | 30
  Change at C3D8; Mean core symptom severity | -0.13 (1.63) | -0.66 (1.20)
  Change at C3D15; Mean core symptom severity: number analyzed (Participants) | 73 | 32
  Change at C3D15; Mean core symptom severity | -0.42 (1.52) | -0.53 (1.05)
  Baseline; Mean module symptom severity: number analyzed (Participants) | 116 | 42
  Baseline; Mean module symptom severity | 1.60 (1.46) | 1.57 (1.11)
  Change at C1D1; Mean module symptom severity: number analyzed (Participants) | 116 | 36
  Change at C1D1; Mean module symptom severity | 0.00 (0.00) | -0.19 (0.96)
  Change at C1D8; Mean module symptom severity: number analyzed (Participants) | 107 | 36
  Change at C1D8; Mean module symptom severity | -0.22 (1.40) | -0.53 (0.96)
  Change at C1D15; Mean module symptom severity: number analyzed (Participants) | 104 | 33
  Change at C1D15; Mean module symptom severity | -0.43 (1.51) | -0.73 (1.13)
  Change at C2D1; Mean module symptom severity: number analyzed (Participants) | 101 | 34
  Change at C2D1; Mean module symptom severity | -0.49 (1.46) | -0.65 (0.92)
  Change at C2D8; Mean module symptom severity: number analyzed (Participants) | 91 | 35
  Change at C2D8; Mean module symptom severity | -0.46 (1.63) | -0.77 (0.87)
  Change at C2D15; Mean module symptom severity: number analyzed (Participants) | 90 | 36
  Change at C2D15; Mean module symptom severity | -0.69 (1.47) | -0.94 (0.93)
  Change at C3D1; Mean module symptom severity: number analyzed (Participants) | 86 | 35
  Change at C3D1; Mean module symptom severity | -0.65 (1.48) | -0.81 (0.97)
  Change at C3D8; Mean module symptom severity: number analyzed (Participants) | 72 | 30
  Change at C3D8; Mean module symptom severity | -0.51 (1.58) | -0.83 (0.97)
  Change at C3D15; Mean module symptom severity: number analyzed (Participants) | 73 | 32
  Change at C3D15; Mean module symptom severity | -0.83 (1.51) | -0.92 (0.97)
  Baseline; Mean interference: number analyzed (Participants) | 116 | 41
  Baseline; Mean interference | 1.81 (2.05) | 1.90 (2.25)
  Change at C1D1; Mean interference: number analyzed (Participants) | 116 | 35
  Change at C1D1; Mean interference | 0.00 (0.00) | -0.13 (1.49)
  Change at C1D8; Mean interference: number analyzed (Participants) | 107 | 33
  Change at C1D8; Mean interference | 0.45 (1.78) | -0.29 (2.14)
  Change at C1D15; Mean interference: number analyzed (Participants) | 104 | 32
  Change at C1D15; Mean interference | 0.36 (1.85) | 0.01 (2.04)
  Change at C2D1; Mean interference: number analyzed (Participants) | 101 | 33
  Change at C2D1; Mean interference | 0.01 (1.73) | -0.34 (1.78)
  Change at C2D8; Mean interference: number analyzed (Participants) | 91 | 34
  Change at C2D8; Mean interference | 0.58 (2.20) | -0.58 (1.81)
  Change at C2D15; Mean interference: number analyzed (Participants) | 89 | 35
  Change at C2D15; Mean interference | 0.06 (1.84) | -0.64 (1.59)
  Change at C3D1; Mean interference: number analyzed (Participants) | 86 | 34
  Change at C3D1; Mean interference | -0.02 (2.02) | -0.73 (2.06)
  Change at C3D8; Mean interference: number analyzed (Participants) | 72 | 29
  Change at C3D8; Mean interference | 0.15 (1.91) | -0.82 (2.09)
  Change at C3D15; Mean interference: number analyzed (Participants) | 72 | 30
  Change at C3D15; Mean interference | -0.07 (2.01) | -0.55 (2.18)

25. Secondary Outcome: Change From Baseline in HRQoL as Measured by European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) Functional Scales Score and Global Health Status/Global Quality-of-Life (QoL) Scale Score
Description: EORTC QLQ-C30 is a validated self-report measure consisting of 30 questions incorporated into 5 functional scales (Physical, Role, Cognitive, Emotional, and Social), 3 symptom scales (fatigue, pain, nausea, and vomiting), a global health status/global QoL scale, and single items (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea). Most questions used 4-point scale (1='Not at all' to 4='Very much'), while 2 questions used 7-point scale (1='very poor' to 7='Excellent'). Scores were averaged, transformed to 0-100 scale; where higher score for functional scales=poor level of functioning; higher score for global health status/global QoL=better HRQoL.
Time Frame: Baseline, D1 of Cycles 1, 2, 3, 4, 5, 6, STC/EW visit (up to C6D28), EoCTR visit (8 to 12 weeks after C6D1), and FUVs (every 12 weeks after EoCTR up to 3 years); Cycle length = 28 days
Population: Patient reported outcome (PRO) evaluable population included all participants with baseline and at least one post-baseline PRO assessment. Here, 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure and 'Number Analyzed' = participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 177 | 69
units on a scale
  Baseline; Physical functioning | 82.59 (17.46) | 83.77 (15.27)
  Change at C1D1; Physical functioning: number analyzed (Participants) | 177 | 67
  Change at C1D1; Physical functioning | 0.0 (0.0) | 1.39 (12.90)
  Change at C2D1; Physical functioning: number analyzed (Participants) | 172 | 67
  Change at C2D1; Physical functioning | 0.31 (15.81) | 2.99 (12.83)
  Change at C3D1; Physical functioning: number analyzed (Participants) | 160 | 64
  Change at C3D1; Physical functioning | 0.22 (16.43) | 1.46 (14.76)
  Change at C4D1; Physical functioning: number analyzed (Participants) | 154 | 65
  Change at C4D1; Physical functioning | 2.11 (14.95) | 5.54 (14.17)
  Change at C5D1; Physical functioning: number analyzed (Participants) | 149 | 65
  Change at C5D1; Physical functioning | 2.44 (18.19) | 4.62 (15.27)
  Change at C6D1; Physical functioning: number analyzed (Participants) | 143 | 65
  Change at C6D1; Physical functioning | 2.25 (16.82) | 4.51 (16.59)
  Change at STC/EW; Physical functioning: number analyzed (Participants) | 162 | 64
  Change at STC/EW; Physical functioning | 1.68 (18.76) | 4.53 (16.04)
  Change at EoCTR; Physical functioning: number analyzed (Participants) | 142 | 63
  Change at EoCTR; Physical functioning | 2.92 (18.03) | 4.34 (16.12)
  Change at FUV1; Physical functioning: number analyzed (Participants) | 124 | 63
  Change at FUV1; Physical functioning | 2.27 (18.86) | 3.81 (16.27)
  Change at FUV2; Physical functioning: number analyzed (Participants) | 114 | 63
  Change at FUV2; Physical functioning | 2.40 (19.21) | 2.75 (17.17)
  Change at FUV3; Physical functioning: number analyzed (Participants) | 95 | 62
  Change at FUV3; Physical functioning | 2.54 (17.83) | 3.44 (17.31)
  Change at FUV4; Physical functioning: number analyzed (Participants) | 77 | 47
  Change at FUV4; Physical functioning | 4.74 (20.14) | 0.85 (21.06)
  Change at FUV5; Physical functioning: number analyzed (Participants) | 57 | 19
  Change at FUV5; Physical functioning | 1.90 (17.68) | -1.75 (19.35)
  Change at FUV6; Physical functioning: number analyzed (Participants) | 33 | 5
  Change at FUV6; Physical functioning | -1.41 (15.34) | 1.33 (5.58)
  Change at FUV7; Physical functioning: number analyzed (Participants) | 13 | 1
  Change at FUV7; Physical functioning | -3.08 (11.74) | 0.00
  Change at FUV8; Physical functioning: number analyzed (Participants) | 5 | 1
  Change at FUV8; Physical functioning | -9.33 (23.38) | 0.00
  Change at FUV9; Physical functioning: number analyzed (Participants) | 2 | 0
  Change at FUV9; Physical functioning | -10.00 (33.0) |
  Baseline; Role functioning | 78.25 (25.67) | 83.82 (21.00)
  Change at C1D1; Role functioning: number analyzed (Participants) | 177 | 67
  Change at C1D1; Role functioning | 0.0 (0.0) | -1.74 (23.23)
  Change at C2D1; Role functioning: number analyzed (Participants) | 172 | 67
  Change at C2D1; Role functioning | -1.26 (27.45) | 2.49 (23.07)
  Change at C3D1; Role functioning: number analyzed (Participants) | 160 | 64
  Change at C3D1; Role functioning | -0.10 (29.64) | 1.82 (26.08)
  Change at C4D1; Role functioning: number analyzed (Participants) | 154 | 65
  Change at C4D1; Role functioning | 0.87 (29.01) | 5.13 (22.03)
  Change at C5D1; Role functioning: number analyzed (Participants) | 149 | 65
  Change at C5D1; Role functioning | 0.45 (30.75) | 4.36 (23.44)
  Change at C6D1; Role functioning: number analyzed (Participants) | 143 | 65
  Change at C6D1; Role functioning | 0.70 (29.92) | 1.79 (25.71)
  Change at STC/EW; Role functioning: number analyzed (Participants) | 162 | 64
  Change at STC/EW; Role functioning | -0.41 (32.91) | 2.60 (25.58)
  Change at EoCTR; Role functioning: number analyzed (Participants) | 143 | 63
  Change at EoCTR; Role functioning | 3.26 (29.95) | 2.12 (26.69)
  Change at FUV1; Role functioning: number analyzed (Participants) | 125 | 63
  Change at FUV1; Role functioning | 2.93 (32.31) | 2.65 (27.47)
  Change at FUV2; Role functioning: number analyzed (Participants) | 114 | 63
  Change at FUV2; Role functioning | 3.07 (32.63) | -1.85 (31.84)
  Change at FUV3; Role functioning: number analyzed (Participants) | 95 | 62
  Change at FUV3; Role functioning | 5.26 (31.16) | 1.88 (28.17)
  Change at FUV4; Role functioning: number analyzed (Participants) | 77 | 47
  Change at FUV4; Role functioning | 5.41 (33.16) | -0.35 (30.39)
  Change at FUV5; Role functioning: number analyzed (Participants) | 57 | 19
  Change at FUV5; Role functioning | 2.34 (29.79) | 1.75 (34.20)
  Change at FUV6; Role functioning: number analyzed (Participants) | 33 | 5
  Change at FUV6; Role functioning | -4.04 (27.01) | -13.33 (32.06)
  Change at FUV7; Role functioning: number analyzed (Participants) | 13 | 1
  Change at FUV7; Role functioning | 2.56 (29.54) | -16.67
  Change at FUV8; Role functioning: number analyzed (Participants) | 5 | 1
  Change at FUV8; Role functioning | 0.00 (23.57) | 16.67
  Change at FUV9; Role functioning: number analyzed (Participants) | 2 | 0
  Change at FUV9; Role functioning | -16.67 (23.57) |
  Baseline; Emotional functioning: number analyzed (Participants) | 176 | 69
  Baseline; Emotional functioning | 78.98 (22.47) | 82.13 (15.80)
  Change at C1D1; Emotional functioning: number analyzed (Participants) | 176 | 67
  Change at C1D1; Emotional functioning | 0.0 (0.0) | 4.35 (15.17)
  Change at C2D1; Emotional functioning: number analyzed (Participants) | 171 | 67
  Change at C2D1; Emotional functioning | 2.24 (20.07) | 5.60 (14.68)
  Change at C3D1; Emotional functioning: number analyzed (Participants) | 158 | 64
  Change at C3D1; Emotional functioning | 2.99 (20.06) | 5.34 (19.09)
  Change at C4D1; Emotional functioning: number analyzed (Participants) | 151 | 65
  Change at C4D1; Emotional functioning | 2.61 (18.35) | 4.19 (15.45)
  Change at C5D1; Emotional functioning: number analyzed (Participants) | 146 | 65
  Change at C5D1; Emotional functioning | 1.14 (18.79) | 3.97 (17.37)
  Change at C6D1; Emotional functioning: number analyzed (Participants) | 143 | 65
  Change at C6D1; Emotional functioning | 2.06 (18.74) | 3.08 (17.96)
  Change at STC/EW; Emotional functioning: number analyzed (Participants) | 160 | 64
  Change at STC/EW; Emotional functioning | 2.43 (20.61) | 5.34 (18.69)
  Change at EoCTR; Emotional functioning: number analyzed (Participants) | 142 | 62
  Change at EoCTR; Emotional functioning | 2.58 (19.45) | 3.49 (17.83)
  Change at FUV1; Emotional functioning: number analyzed (Participants) | 124 | 63
  Change at FUV1; Emotional functioning | 3.49 (20.91) | 4.37 (18.50)
  Change at FUV2; Emotional functioning: number analyzed (Participants) | 114 | 63
  Change at FUV2; Emotional functioning | 4.39 (20.33) | 0.66 (21.02)
  Change at FUV3; Emotional functioning: number analyzed (Participants) | 92 | 62
  Change at FUV3; Emotional functioning | 0.63 (19.97) | 2.82 (17.66)
  Change at FUV4; Emotional functioning: number analyzed (Participants) | 76 | 47
  Change at FUV4; Emotional functioning | 4.82 (19.73) | 1.95 (18.41)
  Change at FUV5; Emotional functioning: number analyzed (Participants) | 56 | 19
  Change at FUV5; Emotional functioning | 3.13 (17.95) | 2.63 (20.61)
  Change at FUV6; Emotional functioning: number analyzed (Participants) | 33 | 5
  Change at FUV6; Emotional functioning | 2.27 (21.78) | 5.00 (17.28)
  Change at FUV7; Emotional functioning: number analyzed (Participants) | 13 | 1
  Change at FUV7; Emotional functioning | 5.77 (17.48) | -8.33
  Change at FUV8; Emotional functioning: number analyzed (Participants) | 5 | 1
  Change at FUV8; Emotional functioning | 3.33 (28.01) | 0.00
  Change at FUV9; Emotional functioning: number analyzed (Participants) | 2 | 0
  Change at FUV9; Emotional functioning | -16.67 (11.79) |
  Baseline; Cognitive functioning: number analyzed (Participants) | 176 | 69
  Baseline; Cognitive functioning | 86.55 (16.78) | 89.86 (14.91)
  Change at C1D1; Cognitive functioning: number analyzed (Participants) | 176 | 67
  Change at C1D1; Cognitive functioning | 0.0 (0.0) | -1.24 (14.01)
  Change at C2D1; Cognitive functioning: number analyzed (Participants) | 171 | 67
  Change at C2D1; Cognitive functioning | -0.19 (15.34) | 0.25 (14.06)
  Change at C3D1; Cognitive functioning: number analyzed (Participants) | 158 | 64
  Change at C3D1; Cognitive functioning | -0.32 (16.34) | -1.56 (17.50)
  Change at C4D1; Cognitive functioning: number analyzed (Participants) | 152 | 65
  Change at C4D1; Cognitive functioning | -1.54 (17.41) | -0.26 (17.05)
  Change at C5D1; Cognitive functioning: number analyzed (Participants) | 146 | 65
  Change at C5D1; Cognitive functioning | -1.94 (18.10) | -0.26 (14.28)
  Change at C6D1; Cognitive functioning: number analyzed (Participants) | 143 | 65
  Change at C6D1; Cognitive functioning | -2.68 (16.97) | -0.77 (15.98)
  Change at STC/EW; Cognitive functioning: number analyzed (Participants) | 160 | 64
  Change at STC/EW; Cognitive functioning | -2.19 (17.65) | 1.04 (18.28)
  Change at EoCTR; Cognitive functioning: number analyzed (Participants) | 142 | 62
  Change at EoCTR; Cognitive functioning | -2.23 (18.11) | -0.27 (16.94)
  Change at FUV1; Cognitive functioning: number analyzed (Participants) | 124 | 63
  Change at FUV1; Cognitive functioning | -2.02 (17.21) | -0.26 (15.98)
  Change at FUV2; Cognitive functioning: number analyzed (Participants) | 114 | 63
  Change at FUV2; Cognitive functioning | 1.32 (16.16) | -2.38 (18.17)
  Change at FUV3; Cognitive functioning: number analyzed (Participants) | 92 | 62
  Change at FUV3; Cognitive functioning | -1.63 (14.84) | -2.96 (18.24)
  Change at FUV4; Cognitive functioning: number analyzed (Participants) | 76 | 47
  Change at FUV4; Cognitive functioning | 0.44 (17.63) | -1.77 (19.11)
  Change at FUV5; Cognitive functioning: number analyzed (Participants) | 56 | 19
  Change at FUV5; Cognitive functioning | -1.49 (15.66) | -6.14 (21.67)
  Change at FUV6; Cognitive functioning: number analyzed (Participants) | 33 | 5
  Change at FUV6; Cognitive functioning | -0.51 (14.72) | 0.00 (0.00)
  Change at FUV7; Cognitive functioning: number analyzed (Participants) | 13 | 1
  Change at FUV7; Cognitive functioning | -1.28 (14.37) | 0.00
  Change at FUV8; Cognitive functioning: number analyzed (Participants) | 5 | 1
  Change at FUV8; Cognitive functioning | 0.00 (23.57) | 0.00
  Change at FUV9; Cognitive functioning: number analyzed (Participants) | 2 | 0
  Change at FUV9; Cognitive functioning | 16.67 (23.57) |
  Baseline; Social functioning: number analyzed (Participants) | 176 | 69
  Baseline; Social functioning | 82.48 (22.06) | 85.51 (21.18)
  Change at C1D1; Social functioning: number analyzed (Participants) | 176 | 67
  Change at C1D1; Social functioning | 0.0 (0.0) | -1.74 (19.92)
  Change at C2D1; Social functioning: number analyzed (Participants) | 171 | 67
  Change at C2D1; Social functioning | -2.44 (21.44) | 0.25 (18.46)
  Change at C3D1; Social functioning: number analyzed (Participants) | 158 | 64
  Change at C3D1; Social functioning | -2.32 (22.61) | 3.65 (25.45)
  Change at C4D1; Social functioning: number analyzed (Participants) | 151 | 65
  Change at C4D1; Social functioning | -0.55 (22.15) | 4.62 (20.09)
  Change at C5D1; Social functioning: number analyzed (Participants) | 146 | 65
  Change at C5D1; Social functioning | -5.48 (26.49) | 2.56 (20.46)
  Change at C6D1; Social functioning: number analyzed (Participants) | 143 | 65
  Change at C6D1; Social functioning | -5.13 (24.80) | 3.85 (24.61)
  Change at STC/EW; Social functioning: number analyzed (Participants) | 160 | 64
  Change at STC/EW; Social functioning | -4.06 (27.71) | 1.04 (19.22)
  Change at EoCTR; Social functioning: number analyzed (Participants) | 142 | 62
  Change at EoCTR; Social functioning | -0.47 (24.95) | 1.88 (20.49)
  Change at FUV1; Social functioning: number analyzed (Participants) | 124 | 63
  Change at FUV1; Social functioning | -1.08 (26.09) | 1.59 (24.27)
  Change at FUV2; Social functioning: number analyzed (Participants) | 114 | 63
  Change at FUV2; Social functioning | 0.58 (24.68) | 1.32 (27.97)
  Change at FUV3; Social functioning: number analyzed (Participants) | 92 | 62
  Change at FUV3; Social functioning | -0.91 (24.00) | 1.88 (25.98)
  Change at FUV4; Social functioning: number analyzed (Participants) | 76 | 47
  Change at FUV4; Social functioning | 1.97 (27.35) | 1.06 (32.12)
  Change at FUV5; Social functioning: number analyzed (Participants) | 56 | 19
  Change at FUV5; Social functioning | 1.79 (26.72) | 0.00 (33.79)
  Change at FUV6; Social functioning: number analyzed (Participants) | 33 | 5
  Change at FUV6; Social functioning | 1.52 (29.27) | 10.00 (14.91)
  Change at FUV7; Social functioning: number analyzed (Participants) | 13 | 1
  Change at FUV7; Social functioning | -2.56 (23.42) | 33.33
  Change at FUV8; Social functioning: number analyzed (Participants) | 5 | 1
  Change at FUV8; Social functioning | -10.00 (22.36) | 33.33
  Change at FUV9; Social functioning: number analyzed (Participants) | 2 | 0
  Change at FUV9; Social functioning | -25.00 (35.36) |
  Baseline; Global health status/QoL: number analyzed (Participants) | 176 | 69
  Baseline; Global health status/QoL | 63.02 (21.45) | 67.39 (22.17)
  Change at C1D1; Global health status/QoL: number analyzed (Participants) | 176 | 67
  Change at C1D1; Global health status/QoL | 0.0 (0.0) | 6.34 (18.41)
  Change at C2D1; Global health status/QoL: number analyzed (Participants) | 171 | 67
  Change at C2D1; Global health status/QoL | 2.73 (21.69) | 5.35 (20.14)
  Change at C3D1; Global health status/QoL: number analyzed (Participants) | 157 | 64
  Change at C3D1; Global health status/QoL | 2.34 (24.66) | 2.21 (23.58)
  Change at C4D1; Global health status/QoL: number analyzed (Participants) | 152 | 65
  Change at C4D1; Global health status/QoL | 3.84 (22.26) | 7.05 (21.05)
  Change at C5D1; Global health status/QoL: number analyzed (Participants) | 146 | 65
  Change at C5D1; Global health status/QoL | 7.36 (24.20) | 7.18 (21.94)
  Change at C6D1; Global health status/QoL: number analyzed (Participants) | 143 | 65
  Change at C6D1; Global health status/QoL | 4.25 (25.00) | 5.90 (25.16)
  Change at STC/EW; Global health status/QoL: number analyzed (Participants) | 160 | 64
  Change at STC/EW; Global health status/QoL | 4.32 (26.20) | 6.51 (23.22)
  Change at EoCTR; Global health status/QoL: number analyzed (Participants) | 142 | 62
  Change at EoCTR; Global health status/QoL | 6.10 (23.65) | 7.66 (24.11)
  Change at FUV1; Global health status/QoL: number analyzed (Participants) | 124 | 63
  Change at FUV1; Global health status/QoL | 5.91 (24.57) | 7.01 (25.01)
  Change at FUV2; Global health status/QoL: number analyzed (Participants) | 114 | 63
  Change at FUV2; Global health status/QoL | 6.94 (24.81) | 4.50 (26.51)
  Change at FUV3; Global health status/QoL: number analyzed (Participants) | 92 | 62
  Change at FUV3; Global health status/QoL | 4.80 (25.30) | 6.32 (27.36)
  Change at FUV4; Global health status/QoL: number analyzed (Participants) | 76 | 47
  Change at FUV4; Global health status/QoL | 7.35 (26.77) | 6.38 (27.60)
  Change at FUV5; Global health status/QoL: number analyzed (Participants) | 56 | 19
  Change at FUV5; Global health status/QoL | 4.46 (23.89) | 4.39 (18.08)
  Change at FUV6; Global health status/QoL: number analyzed (Participants) | 33 | 5
  Change at FUV6; Global health status/QoL | 1.01 (24.00) | 5.00 (7.45)
  Change at FUV7; Global health status/QoL: number analyzed (Participants) | 13 | 1
  Change at FUV7; Global health status/QoL | 8.33 (25.69) | 16.67
  Change at FUV8; Global health status/QoL: number analyzed (Participants) | 5 | 1
  Change at FUV8; Global health status/QoL | 6.67 (16.03) | 8.33
  Change at FUV9; Global health status/QoL: number analyzed (Participants) | 2 | 0
  Change at FUV9; Global health status/QoL | 0.00 (0.00) |

26. Secondary Outcome: Change From Baseline in HRQoL as Measured by Quality of Life Questionnaire Associated CLL Module (QLQ-CLL16) Multi-Item Scales Score
Description: The EORTC QLQ-CLL16 module is designed for participants with Stage 0 to Stage 4 CLL. It is composed of 16 questions and there are four multi-item scales on Fatigue (2 items), Treatment-related side effects (TRSE, 4 items), Disease-related symptoms (DRS, 4 items), and Infection (4 items); and two single-item scales on social activities and future health worries. Multi-item scales score are reported and the total score for each multi-item scale was transformed to result in a total score range of 0 to 100, where higher score = poor HRQoL.
Time Frame: as for outcome 25
Population: PRO evaluable population included all participants with baseline and at least one post-baseline PRO assessment. Here, 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure and 'Number Analyzed' = participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 175 | 69
units on a scale
  Baseline; TRSE | 14.29 (13.95) | 9.42 (8.80)
  Change at C1D1; TRSE: number analyzed (Participants) | 175 | 67
  Change at C1D1; TRSE | 0.0 (0.0) | 0.12 (10.10)
  Change at C2D1; TRSE: number analyzed (Participants) | 170 | 67
  Change at C2D1; TRSE | 1.62 (13.82) | 0.62 (12.76)
  Change at C3D1; TRSE: number analyzed (Participants) | 159 | 63
  Change at C3D1; TRSE | -0.26 (13.76) | 1.98 (14.72)
  Change at C4D1; TRSE: number analyzed (Participants) | 152 | 64
  Change at C4D1; TRSE | -0.49 (13.97) | 0.52 (11.87)
  Change at C5D1; TRSE: number analyzed (Participants) | 147 | 65
  Change at C5D1; TRSE | -0.51 (14.57) | 0.64 (10.02)
  Change at C6D1; TRSE: number analyzed (Participants) | 144 | 65
  Change at C6D1; TRSE | 0.46 (15.51) | -0.13 (10.04)
  Change at STC/EW; TRSE: number analyzed (Participants) | 161 | 64
  Change at STC/EW; TRSE | 0.81 (18.11) | 0.13 (10.76)
  Change at EoCTR; TRSE: number analyzed (Participants) | 142 | 63
  Change at EoCTR; TRSE | -0.88 (16.06) | 0.26 (12.61)
  Change at FUV1; TRSE: number analyzed (Participants) | 123 | 63
  Change at FUV1; TRSE | -1.20 (14.87) | 1.19 (12.24)
  Change at FUV2; TRSE: number analyzed (Participants) | 113 | 63
  Change at FUV2; TRSE | -1.70 (15.28) | 2.65 (14.03)
  Change at FUV3; TRSE: number analyzed (Participants) | 95 | 62
  Change at FUV3; TRSE | -2.08 (12.64) | -0.13 (13.70)
  Change at FUV4; TRSE: number analyzed (Participants) | 76 | 47
  Change at FUV4; TRSE | -1.97 (12.76) | 2.84 (15.18)
  Change at FUV5; TRSE: number analyzed (Participants) | 56 | 19
  Change at FUV5; TRSE | -2.68 (11.02) | 1.32 (10.49)
  Change at FUV6; TRSE: number analyzed (Participants) | 33 | 5
  Change at FUV6; TRSE | -1.01 (12.10) | -1.67 (3.73)
  Change at FUV7; TRSE: number analyzed (Participants) | 13 | 1
  Change at FUV7; TRSE | 2.56 (22.67) | -8.33
  Change at FUV8; TRSE: number analyzed (Participants) | 5 | 1
  Change at FUV8; TRSE | 1.67 (13.69) | 0.00
  Change at FUV9; TRSE: number analyzed (Participants) | 2 | 0
  Change at FUV9; TRSE | 8.33 (11.79) |
  Baseline; DRS | 19.57 (16.81) | 16.95 (17.37)
  Change at C1D1; DRS: number analyzed (Participants) | 175 | 67
  Change at C1D1; DRS | 0.0 (0.0) | -2.74 (16.18)
  Change at C2D1; DRS: number analyzed (Participants) | 170 | 67
  Change at C2D1; DRS | -3.33 (16.05) | -4.77 (16.84)
  Change at C3D1; DRS: number analyzed (Participants) | 159 | 63
  Change at C3D1; DRS | -4.77 (16.49) | -3.35 (17.48)
  Change at C4D1; DRS: number analyzed (Participants) | 152 | 64
  Change at C4D1; DRS | -6.03 (16.51) | -5.12 (17.72)
  Change at C5D1; DRS: number analyzed (Participants) | 147 | 65
  Change at C5D1; DRS | -5.90 (16.73) | -4.79 (17.50)
  Change at C6D1; DRS: number analyzed (Participants) | 144 | 65
  Change at C6D1; DRS | -6.40 (17.26) | -5.30 (16.72)
  Change at STC/EW; DRS: number analyzed (Participants) | 161 | 64
  Change at STC/EW; DRS | -5.80 (18.52) | -6.51 (18.45)
  Change at EoCTR; DRS: number analyzed (Participants) | 142 | 63
  Change at EoCTR; DRS | -6.57 (17.21) | -5.86 (20.38)
  Change at FUV1; DRS: number analyzed (Participants) | 123 | 63
  Change at FUV1; DRS | -6.55 (15.73) | -5.82 (19.20)
  Change at FUV2; DRS: number analyzed (Participants) | 113 | 63
  Change at FUV2; DRS | -8.63 (14.39) | -3.57 (18.31)
  Change at FUV3; DRS: number analyzed (Participants) | 95 | 62
  Change at FUV3; DRS | -7.37 (14.88) | -3.76 (19.25)
  Change at FUV4; DRS: number analyzed (Participants) | 76 | 47
  Change at FUV4; DRS | -8.55 (18.56) | -2.66 (20.49)
  Change at FUV5; DRS: number analyzed (Participants) | 56 | 19
  Change at FUV5; DRS | -8.33 (16.13) | -2.19 (19.41)
  Change at FUV6; DRS: number analyzed (Participants) | 33 | 5
  Change at FUV6; DRS | -6.31 (16.01) | -3.33 (13.94)
  Change at FUV7; DRS: number analyzed (Participants) | 13 | 1
  Change at FUV7; DRS | -15.38 (20.08) | -8.33
  Change at FUV8; DRS: number analyzed (Participants) | 5 | 1
  Change at FUV8; DRS | -10.00 (16.03) | -8.33
  Change at FUV9; DRS: number analyzed (Participants) | 2 | 0
  Change at FUV9; DRS | -4.17 (5.89) |
  Baseline; Fatigue | 28.76 (24.66) | 21.74 (20.67)
  Change at C1D1; Fatigue: number analyzed (Participants) | 175 | 67
  Change at C1D1; Fatigue | 0.0 (0.0) | -2.24 (20.29)
  Change at C2D1; Fatigue: number analyzed (Participants) | 170 | 67
  Change at C2D1; Fatigue | -2.55 (22.86) | -5.47 (21.40)
  Change at C3D1; Fatigue: number analyzed (Participants) | 159 | 63
  Change at C3D1; Fatigue | -2.83 (25.17) | -3.17 (23.73)
  Change at C4D1; Fatigue: number analyzed (Participants) | 152 | 64
  Change at C4D1; Fatigue | -3.18 (23.23) | -4.17 (22.02)
  Change at C5D1; Fatigue: number analyzed (Participants) | 147 | 65
  Change at C5D1; Fatigue | -2.38 (27.52) | -4.36 (20.89)
  Change at C6D1; Fatigue: number analyzed (Participants) | 144 | 65
  Change at C6D1; Fatigue | -2.66 (26.35) | -2.31 (21.42)
  Change at STC/EW; Fatigue: number analyzed (Participants) | 161 | 64
  Change at STC/EW; Fatigue | -3.11 (28.64) | -4.69 (21.30)
  Change at EoCTR; Fatigue: number analyzed (Participants) | 142 | 63
  Change at EoCTR; Fatigue | -6.69 (26.78) | -3.97 (24.27)
  Change at FUV1; Fatigue: number analyzed (Participants) | 123 | 63
  Change at FUV1; Fatigue | -6.37 (26.61) | -4.23 (22.99)
  Change at FUV2; Fatigue: number analyzed (Participants) | 113 | 63
  Change at FUV2; Fatigue | -6.64 (24.55) | -1.85 (24.70)
  Change at FUV3; Fatigue: number analyzed (Participants) | 95 | 62
  Change at FUV3; Fatigue | -5.79 (23.29) | -2.42 (23.73)
  Change at FUV4; Fatigue: number analyzed (Participants) | 76 | 47
  Change at FUV4; Fatigue | -9.65 (26.84) | -0.35 (25.18)
  Change at FUV5; Fatigue: number analyzed (Participants) | 56 | 19
  Change at FUV5; Fatigue | -6.55 (25.56) | 3.51 (23.95)
  Change at FUV6; Fatigue: number analyzed (Participants) | 33 | 5
  Change at FUV6; Fatigue | -5.05 (24.82) | 3.33 (24.72)
  Change at FUV7; Fatigue: number analyzed (Participants) | 13 | 1
  Change at FUV7; Fatigue | -10.26 (30.08) | -33.33
  Change at FUV8; Fatigue: number analyzed (Participants) | 5 | 1
  Change at FUV8; Fatigue | -6.67 (19.00) | 0.00
  Change at FUV9; Fatigue: number analyzed (Participants) | 2 | 0
  Change at FUV9; Fatigue | -8.33 (11.79) |
  Baseline; Infection | 15.92 (17.63) | 14.01 (18.99)
  Change at C1D1; Infection: number analyzed (Participants) | 175 | 67
  Change at C1D1; Infection | 0.0 (0.0) | -2.24 (20.03)
  Change at C2D1; Infection: number analyzed (Participants) | 170 | 67
  Change at C2D1; Infection | -0.02 (19.98) | -3.61 (21.72)
  Change at C3D1; Infection: number analyzed (Participants) | 159 | 63
  Change at C3D1; Infection | -1.66 (19.21) | -1.32 (20.48)
  Change at C4D1; Infection: number analyzed (Participants) | 152 | 64
  Change at C4D1; Infection | -1.44 (22.07) | -3.13 (21.28)
  Change at C5D1; Infection: number analyzed (Participants) | 147 | 65
  Change at C5D1; Infection | -1.91 (24.00) | -2.56 (23.47)
  Change at C6D1; Infection: number analyzed (Participants) | 143 | 65
  Change at C6D1; Infection | -1.09 (20.66) | -2.95 (20.54)
  Change at STC/EW; Infection: number analyzed (Participants) | 161 | 64
  Change at STC/EW; Infection | -0.12 (23.28) | -1.69 (23.34)
  Change at EoCTR; Infection: number analyzed (Participants) | 142 | 63
  Change at EoCTR; Infection | -0.55 (21.73) | -3.44 (25.78)
  Change at FUV1; Infection: number analyzed (Participants) | 121 | 63
  Change at FUV1; Infection | 1.08 (18.77) | -2.65 (26.51)
  Change at FUV2; Infection: number analyzed (Participants) | 113 | 63
  Change at FUV2; Infection | 0.05 (23.29) | -0.53 (25.74)
  Change at FUV3; Infection: number analyzed (Participants) | 95 | 62
  Change at FUV3; Infection | -1.90 (16.97) | -0.54 (26.48)
  Change at FUV4; Infection: number analyzed (Participants) | 76 | 47
  Change at FUV4; Infection | -4.24 (16.71) | 0.53 (25.56)
  Change at FUV5; Infection: number analyzed (Participants) | 56 | 19
  Change at FUV5; Infection | -4.51 (22.66) | 7.46 (27.20)
  Change at FUV6; Infection: number analyzed (Participants) | 33 | 5
  Change at FUV6; Infection | -1.60 (18.90) | 8.33 (15.59)
  Change at FUV7; Infection: number analyzed (Participants) | 13 | 1
  Change at FUV7; Infection | -0.43 (21.84) | -16.67
  Change at FUV8; Infection: number analyzed (Participants) | 5 | 1
  Change at FUV8; Infection | 8.89 (23.36) | -25.00
  Change at FUV9; Infection: number analyzed (Participants) | 2 | 0
  Change at FUV9; Infection | -2.78 (3.93) |

27. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered with Mircera and which does not necessarily have a causal relationship with Mircera. A Serious Adverse Event (SAE) is any significant hazard, contraindication, side effect that is fatal or life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is medically significant or requires intervention to prevent one or other of the outcomes listed above. AEs were assessed using National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE, v4.0)
Time Frame: From signing of informed consent form up to approximately 8 years 5 months
Population: SE population included all randomized participants who received at least one dose of study treatment with participants grouped according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 188 | 194
Participants
  Adverse Events | 185 | 194
  Serious Adverse Events | 84 | 101

28. Secondary Outcome: Number of Participants With Grade 3 or Higher Tumor Lysis Syndrome (TLS) and Infusion-related Reactions (IRRs)
Description: An AE was defined as any untoward medical occurrence in a participant administered with Mircera and which does not necessarily have a causal relationship with Mircera. A SAE is any significant hazard, contraindication, side effect that is fatal or life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is medically significant or requires intervention to prevent one or other of the outcomes listed above. TLS and IRRs were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant; Grade 4 = Life-threatening; Grade 5 = Death. A higher grade indicates a worse outcome.
Time Frame: From signing of informed consent form up to approximately 8 years 5 months
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study
Number analyzed (Participants) | 188 | 194
Participants
  TLS | 2 | 6
  IRRs | 10 | 4

29. Other Pre Specified Outcome: Change From Baseline in Lymphocyte Subset Counts at Specified Time Points
Time Frame: Baseline, C4D14-28, Study Treatment Completion/Early Withdrawal (STC/EW, up to C6D28), EoCTR visit (8 to 12 weeks after C6D1), and at FUVs (every 12 weeks after EoCTR up to 3 years); Cycle length = 28 days
Reporting Status: Not Posted

30. Post Hoc Outcome: Euro QoL 5 Dimension (EQ-5D) Questionnaire Score
Time Frame: as for outcome 25
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From signing of informed consent form up to approximately 8 years 5 months
Description: SE population included all randomized participants who received at least one dose of study treatment with participants grouped according to the actual treatment received.
Groups:
- Bendamustine + Rituximab Main Study: Participants received bendamustine at a dose of 70 mg/m^2 via IV infusion on Days 1 and 2 of each 28-day cycle for 6 cycles, in combination with rituximab at a dose of 375 mg/m^2 via IV infusion on Day 1 of Cycle 1 and at a dose of 500 mg/m^2 on Day 1 of Cycles 2-6.
- Venetoclax + Rituximab Main Study: Participants were initially placed on a venetoclax ramp-up period of 5 weeks, and received an initial dose of 20 mg via tablet orally QD for initial 1 to 7 days, then venetoclax dose was incremented weekly up to a maximum dose of 400 mg via tablet orally QD. Participants continued receiving venetoclax at a dose of 400 mg via tablet orally QD from Week 6 (Day 1 of Cycle 1 of combination therapy) onwards up to PD or 2 years, whichever occurred first, as directed by the investigator, in combination with rituximab at a dose of 375 mg/m^2 via IV infusion on Day 1 of Cycle 1 and at a dose of 500 mg/m^2 on Day 1 of Cycles 2-6.
Arm/Group | Bendamustine + Rituximab Main Study | Venetoclax + Rituximab Main Study | Bendamustine + Rituximab Crossover Substudy | Venetoclax + Rituximab Re-Treatment Substudy
All-Cause Mortality (participants affected / at risk) | 84/188 | 60/194 | 1/9 | 8/25
Serious Adverse Events (participants affected / at risk) | 84/188 | 101/194 | 5/9 | 13/25
Other Adverse Events (participants affected / at risk) | 177/188 | 190/194 | 5/9 | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine + Rituximab Main Study (N=188) | Venetoclax + Rituximab Main Study (N=194) | Bendamustine + Rituximab Crossover Substudy (N=9) | Venetoclax + Rituximab Re-Treatment Substudy (N=25)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 3 (4) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (16) | 7 (7) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (4) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Listeria sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Moraxella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritoneal tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 15 (17) | 19 (23) | 1 (2) | 3 (4)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Scedosporium infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 6 (8) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperpyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 13 (15) | 5 (5) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical observation (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sebaceous adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (7) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine + Rituximab Main Study (N=188) | Venetoclax + Rituximab Main Study (N=194) | Bendamustine + Rituximab Crossover Substudy (N=9) | Venetoclax + Rituximab Re-Treatment Substudy (N=25)
Anaemia (Blood and lymphatic system disorders) | 40 (68) | 28 (48) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 84 (182) | 120 (290) | 3 (5) | 5 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 42 (57) | 23 (30) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 13 (14) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 39 (47) | 27 (31) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 31 (43) | 78 (120) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 64 (82) | 42 (58) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 22 (29) | 15 (18) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 13 (14) | 20 (32) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 5 (5) | 10 (11) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 11 (15) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (15) | 22 (29) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 12 (12) | 8 (11) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 14 (17) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5) | 19 (26) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 28 (42) | 45 (81) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 7 (9) | 12 (22) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 40 (54) | 16 (21) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 10 (11) | 10 (17) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 13 (27) | 11 (27) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 17 (18) | 8 (11) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 11 (16) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 11 (12) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (15) | 17 (22) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 14 (14) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (11) | 4 (4) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 11 (14) | 12 (14) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 19 (21) | 21 (21) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 12 (13) | 21 (22) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (37) | 36 (51) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 11 (14) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (12) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 12 (14) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 10 (11) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 25 (29) | 15 (19) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 15 (15) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 16 (20) | 8 (10) | 0 (0) | 1 (1)
Fatigue (General disorders) | 39 (44) | 35 (41) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 7 (11) | 10 (14) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 33 (44) | 27 (41) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 5 (6) | 1 (2) | 0 (0)
White blood cell count decreased (Investigations) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT02005471/Prot_002.pdf
  • Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT02005471/SAP_001.pdf